CLINICAL TRIAL: NCT03390296
Title: An Open-Label Phase Ib/II Multi-Arm Study of OX40 Agonist Monoclonal Antibody (mAb), Anti-PDL1 mAb, Smoothened Inhibitor, Anti-CD33 mAb, Bcl-2 Inhibitor and Azacitidine as Single-Agents and/or Combinations for the Treatment of Patients With Acute Myeloid Leukemia (AML)
Brief Title: OX40, Venetoclax, Avelumab, Glasdegib, Gemtuzumab Ozogamicin, and Azacitidine in Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0337; NCI-2018-00972 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0337 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — avelumab; Azacitidine; Gemtuzumab; glasdegib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (anti-OX40 antibody PF-04518600) (Experimental): Patients receive anti-OX40 antibody PF-04518600 IV over 60 minutes on days 1 and 14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-OX40 Agonist Monoclonal Antibody PF-04518600
- Arm B (azacitidine, venetoclax, GO) (Experimental): Patients receive azacitidine IV over 10-40 minutes or via injection SC on days 1-7 or 1-5 and 8-9. Patients also receive venetoclax PO on days 1-28 and GO IV over 2 hours on day 8. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Gemtuzumab Ozogamicin; Drug: Venetoclax
- Arm C (azacitidine, GO, avelumab) (Experimental): Patients receive azacitidine and GO as in Arm B. Patients also receive avelumab IV over 60 minutes on days 1 and 14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Gemtuzumab Ozogamicin; Drug: Azacitidine
- Arm D (azacitidine, venetoclax, avelumab) (Experimental): Patients receive azacitidine and venetoclax as in Arm A and avelumab as in Arm C. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Azacitidine; Drug: Venetoclax
- Arm E (azacitidine, avelumab, anti-OX40 antibody PF-04518600) (Experimental): Patients receive azacitidine and avelumab as in Arm C and anti-OX40 antibody PF-04518600 as in Arm A. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-OX40 Agonist Monoclonal Antibody PF-04518600; Drug: Avelumab; Drug: Azacitidine
- Arm F (GO, glasdegib) (Experimental): Patients receive GO IV over 2 hours on days 1, 4, and 7, and glasdegib PO on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemtuzumab Ozogamicin; Drug: Glasdegib; Drug: Glasdegib Maleate

INTERVENTIONS:
Biological: Anti-OX40 Agonist Monoclonal Antibody PF-04518600 — Given IV
  Other Names: PF-04518600; PF04518600
  Arms: Arm A (anti-OX40 antibody PF-04518600); Arm E (azacitidine, avelumab, anti-OX40 antibody PF-04518600)
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
  Arms: Arm C (azacitidine, GO, avelumab); Arm D (azacitidine, venetoclax, avelumab); Arm E (azacitidine, avelumab, anti-OX40 antibody PF-04518600)
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm B (azacitidine, venetoclax, GO); Arm D (azacitidine, venetoclax, avelumab); Arm E (azacitidine, avelumab, anti-OX40 antibody PF-04518600)
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
  Arms: Arm B (azacitidine, venetoclax, GO); Arm C (azacitidine, GO, avelumab); Arm F (GO, glasdegib)
Drug: Glasdegib — Given PO
  Other Names: PF 04449913; PF-04449913; PF04449913
  Arms: Arm F (GO, glasdegib)
Drug: Glasdegib Maleate — Given PO
  Other Names: Daurismo; PF 04449913 Maleate
  Arms: Arm F (GO, glasdegib)
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
  Arms: Arm B (azacitidine, venetoclax, GO); Arm D (azacitidine, venetoclax, avelumab)
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496
  Arms: Arm C (azacitidine, GO, avelumab)

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of anti-OX40 antibody PF-04518600 (OX40) and how well it works alone or in combination with venetoclax, avelumab, glasdegib, gemtuzumab ozogamicin, and azacitidine in treating patients with acute myeloid leukemia that has come back or does not respond to treatment. Immunotherapy with monoclonal antibodies, such as OX40, avelumab, and gemtuzumab ozogamicin, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Glasdegib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as venetoclax and azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving OX40, venetoclax, avelumab, glasdegib, gemtuzumab ozogamicin, and azacitidine may work better in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of multiple combination regimens of IO-agents (PF04518600 [Ox40 agonist monoclonal antibody (mAb)], avelumab [PD-L1 antagonist mAb], hypomethylator therapy (azacitidine), anti CD33 mAb (gemtuzumab ozogamycin, GO), Bcl-2 inhibitor (venetoclax) and smoothened pathway inhibitor (glasdegib) in patients with relapsed/refractory (RR) acute myeloid leukemia (AML).

II. To evaluate the composite complete response (CRc) defined as complete response (CR) + complete response with incomplete recovery of platelets (CRp) + complete response with incomplete recovery of counts (CRi) within 3 months of therapy initiation in patients with RR AML of: Arm A. PF-04518600 alone, Arm B. azacitidine + venetoclax + GO, Arm C. azacitidine + aveluma + GO, Arm D. azacitidine + venetoclax + avelumab, Arm E. Azacitidine + avelumab + PF-04518600, Arm F. GO + glasdegib.

SECONDARY OBJECTIVES:

I. To assess the morphologic leukemia free survival (MLFS), partial response (PR), hematologic improvement (HI) rate of patients with RR AML treated on arms A-F.

II. To assess relapse-free survival (RFS), time to next therapy (TNT), 4-week and 8-week mortality, and overall survival (OS) of patients with RR AML treated on arms A-F.

III. To assess minimal residual disease (MRD) by multiparametric flow-cytometry at response (+/- 1 month) and assess correlation of MRD to OS in arms A-F.

EXPLORATORY OBJECTIVES:

I. To study immunological and molecular features at baseline and at predefined time-points on-therapy with each combination in the peripheral blood and bone marrow to include quantification of immune ligand expression by the AML/myelodysplastic syndrome (MDS) blasts and AML/MDS stromal components (myeloid-derived suppressor cell [MDSC]s, monocytes and mesenchymal stem cell [MSC]s) including galectin 9, 4-1BBL, ICOSL, PD-L1, PD-L2, OX-40L, CD137L, others.

II. To study immunological and molecular features at baseline and at predefined time-points on-therapy with each combination in the peripheral blood and bone marrow to include determination of the quantitative expression of positive and negative co-stimulatory molecules including 4-1BB, CTLA-4, ICOS, PD-1, OX40, LAG-3, TIM-3, HLA-DR, Ki67, others on T-lymphocyte subsets.

III. To study immunological and molecular features at baseline and at predefined time-points on-therapy with each combination in the peripheral blood and bone marrow to include identification of the immunophenotype of tumor-infiltrating T-lymphocytes (TILs) pre- and post-therapy including CD8+, CD4+ effector, CD4+ regulatory TILs and central memory, effector memory, and naive T-cell subsets among the CD4 and CD8 populations.

IV. To develop a micro-array based gene expression profile (GEP) predictor of response to the immune combinations using either baseline ribonucleic acid (RNA) sequencing and/or nanostring.

V. To perform a validated next generation sequencing (NGS)-based analysis for the detection of somatic mutations in the coding sequences of 28 genes commonly mutated in AML at baseline and on treatment to identify baseline predictors and clonal evolution on treatment and/or whole exome sequencing (WES) in selected cases.

VI. To identify clonal T-cells by performing T-cell repertoire analysis at baseline and longitudinally on therapy on the peripheral blood and/o bone marrow samples.

VII. To assess levels of cytokines at baseline and longitudinally on therapy in peripheral blood and/or bone marrow.

OUTLINE: This is a phase I, dose escalation study of anti-OX40 antibody PF-04518600 followed by a phase II study. Patients are assigned to 1 of 6 arms.

ARM A: Patients receive anti-OX40 antibody PF-04518600 intravenously (IV) over 60 minutes on days 1 and 14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive azacitidine IV over 10-40 minutes or via injection subcutaneously (SC) on days 1-7 or 1-5 and 8-9. Patients also receive venetoclax orally (PO) on days 1-28 and GO IV over 2 hours on day 8. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive azacitidine and GO as in Arm B. Patients also receive avelumab IV over 60 minutes on days 1 and 14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive azacitidine and venetoclax as in Arm A and avelumab as in Arm C. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM E: Patientss receive azacitidine and avelumab as in Arm C and anti-OX40 antibody PF-04518600 as in Arm A. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM F: Patients receive GO IV over 2 hours on days 1, 4, and 7, and glasdegib PO on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After conclusion of study treatment, patients are followed up at 30 days, then every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* ARMS A-G: RR AML: Patients with AML who are refractory or relapsed (any salvage) with no available therapies or not candidates for available therapies. For patients with prior MDS or chronic myelomonocytic leukemia (CMML) or myeloproliferative neoplasm (MPN) who transformed to AML, therapy received for MDS, CMML, or MPN is NOT considered as prior therapy for AML with the exception of MDS or CMML treated with hypomethylating agents (HMAs). Patients with MDS or CMML treated with HMA therapies who progress to AML, and have no available therapies or are not candidates for available therapies, will be eligible at the time of progression to AML.
* Prior therapy with hydroxyurea, chemotherapy, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Total bilirubin =< 2.0 times upper limit of normal (x ULN).
* Aspartate aminotransferase or alanine aminotransferase =< 2.5 x ULN (aspartate aminotransferase or alanine aminotransferase =< 5.0 x ULN if deemed related to leukemia by the treating physician).
* Adequate renal function defined by an estimated creatinine clearance >= 40 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
* Patients must provide written informed consent.
* In the absence of rapidly progressive disease, the interval from prior treatment to the time of initiation of protocol therapy will be at least 14 days for prior anti-leukemic therapy, with the exception of hydroxyurea as noted below, OR at least 5 half-lives for cytotoxic/noncytotoxic agents, whichever is shorter. The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochure's, or drug-administration manuals) and will be documented in the protocol eligibility document. The toxicity from prior therapy should have resolved to grade =< 1, however alopecia and sensory neuropathy grade =< 2 not constituting a safety risk based on investigators judgement is acceptable. Since the effect of most IO-agents, HMA-therapies, SMO-inhibitors, venetoclax may be delayed, use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and will not require a washout.
* Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted. Patients with a known history of CNS disease or leukemic brain metastasis must have been treated locally, have at least 3 consecutive lumbar punctures (LPs) with no evidence of CNS leukemia, and must be clinically stable for at least 4 weeks prior to enrollment and have no ongoing neurological symptoms that in the opinion of the treating physician are related to the CNS disease (sequelae that are a consequence of the treatment of the CNS disease are acceptable).
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment.
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment. Adequate methods of contraception include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient.
  * Combination of any of the two following:

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository in case of use of oral contraception, women should have been stable on the same pill before taking study treatment.
  * Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Exclusion Criteria:

* Patients with a known allergy or hypersensitivity to the protocol therapies or any of their components to be used in the arm the patient is to be enrolled on. Known severe hypersensitivity reactions to monoclonal antibodies (grade >= 3 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
* Patients with a known history of severe interstitial lung disease or severe pneumonitis or active pneumonitis/pneumonia or pulmonary pathology that is not well controlled in the opinion of the treating physician and/or principal investigator (PI).
* Clinically significant (i.e., active) cardiovascular disease: acute cerebral vascular accident/stroke (< 6 months prior to enrollment) excluding transient ischemic attack (TIA), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association classification class II), or serious cardiac arrhythmia requiring medication.
* Ejection fraction < 50% on screening echocardiography (ECHO) or multigated acquisition scan (MUGA).
* Persisting toxicity related to prior therapy of grade > 1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy grade =< 2 is acceptable.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent: * Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible

  * Current use of immunosuppressive medication, EXCEPT for the following:

    * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
    * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent;
    * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).
* Prior organ transplantation including allogenic stem-cell transplantation within 3 months prior to planned enrollment.
* Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia.
* Active and uncontrolled disease (active infection requiring systemic therapy, fever likely secondary to infection within prior 48 hours, uncontrolled hypertension despite adequate medical therapy as judged by the treating physician.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive.
* Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
* Other severe acute or chronic medical conditions that is active and not well controlled including colitis, inflammatory bowel disease, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Patients unwilling or unable to comply with the protocol.
* Pregnant or breastfeeding.
* Known alcohol or drug abuse within the last 1 year.
* Acute promyelocytic leukemia (APL).
* Cardiac exclusions specific to glasdegib and OX40 containing arms: Any one of the following ongoing or in the previous 6 months: congenital long QT syndrome, torsades de pointes or any clinically significant ventricular fibrillation, sustained ventricular tachyarrhythmia requiring medical intervention, right bundle branch block + left anterior hemiblock (i.e. bifascicular block): isolated RBBB without a bifascicular block will not be an exclusion criterion; complete left bundle branch block, unstable angina or myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident (CVA), transient ischemic attack or symptomatic pulmonary emboli, as well as bradycardia defined as < 50 bpms on screening or day 1 electrocardiography (EKG). Known history of second or third degree heart block (may be eligible if the patient currently has a pacemaker). Active cardiac dysrhythmias of NCI CTCAE grade >= 2 (eg, atrial fibrillation) or corrected QT interval by Fridericia's correction formula (QTcF) interval > 470 msec within 4 weeks prior to starting the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval G Daver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Short NJ, Borthakur G, Pemmaraju N, Dinardo CD, Kadia TM, Jabbour E, Konopleva M, Macaron W, Ning J, Ma J, Pierce S, Alvarado Y, Sasaki K, Takahashi K, Estrov Z, Masarova L, Issa GC, Montalban-Bravo G, Andreeff M, Burger JA, Miller D, Alexander L, Naing A, Garcia-Manero G, Ravandi F, Daver N. A multi-arm phase Ib/II study designed for rapid, parallel evaluation of novel immunotherapy combinations in relapsed/refractory acute myeloid leukemia. Leuk Lymphoma. 2022 Sep;63(9):2161-2170. doi: 10.1080/10428194.2022.2062345. Epub 2022 Apr 20. PMID 35442137
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Zero participants were registered on Arm E.
Period: Overall Study
Arm/Group | Arm A (Anti-OX40 Antibody PF-04518600) | Arm B (Azacitidine, Venetoclax, GO) | Arm C (Azacitidine, GO, Avelumab) | Arm D (Azacitidine, Venetoclax, Avelumab) | Arm E (Azacitidine, Avelumab, Anti-OX40 Antibody PF-04518600) | Arm F (GO, Glasdegib)
Started | 4 | 21 | 7 | 13 | 0 | 5
Completed | 4 | 21 | 7 | 13 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero participants were registered on Arm E.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Anti-OX40 Antibody PF-04518600) | Arm B (Azacitidine, Venetoclax, GO) | Arm C (Azacitidine, GO, Avelumab) | Arm D (Azacitidine, Venetoclax, Avelumab) | Arm E (Azacitidine, Avelumab, Anti-OX40 Antibody PF-04518600) | Arm F (GO, Glasdegib) | Total
Number analyzed (Participants) | 4 | 21 | 7 | 13 | 0 | 5 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Between 18 and 65 years | 3 | 10 | 4 | 5 | 0 | 2 | 24
  >=65 years | 0 | 11 | 3 | 8 | 0 | 2 | 24
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 62] | 66 [27 to 84] | 63 [29 to 79] | 67 [47 to 73] |  | 64 [18 to 67] | 64 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 10 | 4 | 5 |  | 3 | 23
  Male | 3 | 11 | 3 | 8 |  | 2 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 |  | 0 | 0
  Asian | 0 | 1 | 0 | 0 |  | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 |  | 1 | 4
  White | 3 | 17 | 6 | 11 |  | 4 | 41
  More than one race | 0 | 0 | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 0 | 3 | 1 | 0 |  | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 21 | 7 | 13 |  | 5 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: Response is: CR + complete response with incomplete recovery of platelets (CRp) + complete response with incomplete recovery of counts (CRi) within 3 months. CR: Bone Marrow blasts </= 5%, Absolute neutrophil count >/= 1,000, Platelets >/= 100 and no extra medullary disease.CRp: Bone Marrow blasts </= 5%, Absolute neutrophil count >/= 1,000 and no extra medullary disease. CRi: Bone Marrow blasts </= 5%
Time Frame: within 3 months of initiation of therapy
Population: Zero participants were registered on Arm E. Four participants in Arm B, One participant in arm C, two participants in arm D and two participants in arm F were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Anti-OX40 Antibody PF-04518600) | Arm B (Azacitidine, Venetoclax, GO) | Arm C (Azacitidine, GO, Avelumab) | Arm D (Azacitidine, Venetoclax, Avelumab) | Arm E (Azacitidine, Avelumab, Anti-OX40 Antibody PF-04518600) | Arm F (GO, Glasdegib)
Number analyzed (Participants) | 4 | 17 | 6 | 11 | 0 | 3
Participants | 0 | 8 | 1 | 2 |  | 0

2. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A (Anti-OX40 Antibody PF-04518600) | Arm B (Azacitidine, Venetoclax, GO) | Arm C (Azacitidine, GO, Avelumab) | Arm D (Azacitidine, Venetoclax, Avelumab) | Arm E (Azacitidine, Avelumab, Anti-OX40 Antibody PF-04518600) | Arm F (GO, Glasdegib)
Number analyzed (Participants) | 4 | 17 | 6 | 11 | 0 | 3
Months | 3.0 [2.5 to 17.9] | 7.6 [0.7 to 30.3] | 5.9 [2.9 to 37.7] | 4.8 [1.0 to 34.0] |  | 1.1 [0.3 to 1.8]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Zero participants were registered on Arm E.
Arm/Group | Arm A (Anti-OX40 Antibody PF-04518600) | Arm B (Azacitidine, Venetoclax, GO) | Arm C (Azacitidine, GO, Avelumab) | Arm D (Azacitidine, Venetoclax, Avelumab) | Arm E (Azacitidine, Avelumab, Anti-OX40 Antibody PF-04518600) | Arm F (GO, Glasdegib)
All-Cause Mortality (participants affected / at risk) | 1/4 | 3/21 | 1/7 | 2/13 | 0/0 | 5/5
Serious Adverse Events (participants affected / at risk) | 3/4 | 17/21 | 6/7 | 9/13 | 0/0 | 5/5
Other Adverse Events (participants affected / at risk) | 3/4 | 5/21 | 1/7 | 3/13 | 0/0 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Anti-OX40 Antibody PF-04518600) (N=4) | Arm B (Azacitidine, Venetoclax, GO) (N=21) | Arm C (Azacitidine, GO, Avelumab) (N=7) | Arm D (Azacitidine, Venetoclax, Avelumab) (N=13) | Arm E (Azacitidine, Avelumab, Anti-OX40 Antibody PF-04518600) (N=0) | Arm F (GO, Glasdegib) (N=5)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 7 (10) | 2 (4) | 3 (3) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune System Disorders (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 6 (10) | 3 (3) | 3 (7) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha Hemolytic Strep Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
septicemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Anti-OX40 Antibody PF-04518600) (N=4) | Arm B (Azacitidine, Venetoclax, GO) (N=21) | Arm C (Azacitidine, GO, Avelumab) (N=7) | Arm D (Azacitidine, Venetoclax, Avelumab) (N=13) | Arm E (Azacitidine, Avelumab, Anti-OX40 Antibody PF-04518600) (N=0) | Arm F (GO, Glasdegib) (N=5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03390296/Prot_SAP_000.pdf